CLINICAL TRIAL: NCT06515145
Title: To Evaluate the Safety and Efficacy of High-volume Versus Standard Volume Plasma Exchange in Patients With Acute Liver Failure With Cerebral Edema -A Prospective Randomized Controlled Trial
Brief Title: High-volume Versus Standard Volume Plasma Exchange in Patients With Acute Liver Failure With Cerebral Edema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALFCE-01
Record Dates: First submitted 2024-06-18; First posted 2024-07-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Liver Failure; Cerebral Edema
Keywords: Plasma-exchange; systemic inflammatory response syndrome; lactate; CRRT; sepsis
MeSH Terms: conditions — Liver Failure, Acute; Brain Edema; Systemic Inflammatory Response Syndrome; Sepsis

STUDY DESIGN:
Intervention Model Description: Intervention : High Volume Therapeutic Plasma Exchange (HVPE)+ Standard Medical Treatment (SMT) The high-volume strategy would be performed by centrifugation technique ~ 8-9 litres of plasma would be exchanged in each patient over 6-8 hours.
  Active Comparator - The Standard volume Plasma Exchange + Standard medical Treatment The Standard volume strategy group Therapeutic Plasma Exchange would be performed varying from 1.5- 2.5 times the plasma - volume.
Masking Description: As it is a Medicinal intervention masking of the either of participants or investigator or other investigator is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Volume Therapeutic plasma Exchange (Experimental): The high - volume strategy would be performed by centrifugation technique ~ 8 - 9 litres of plasma would be exchanged in each patient over 6 - 8 hours along with Standard Medical Treatment
  Interventions: Procedure: High Volume Therapeutic Plasma Exchange
- Standard volume Therapeutic Plasma Exchange (Active Comparator): The standard volume strategy would be performed centrifugation technique with Plasma volume varying from 1.5 - 2.5 times the plasma - volume along with Standard Medical Treatment.
  Interventions: Procedure: Standard volume therapeutic plasma exchange

INTERVENTIONS:
Procedure: High Volume Therapeutic Plasma Exchange — Experimental- High Volume Therapeutic Plasma Exchange at (8 - 9 litres of plasma would be exchanged in each patient over 6 - 8 hours)
  Arms: High Volume Therapeutic plasma Exchange
Procedure: Standard volume therapeutic plasma exchange — Active Comparator - The standard volume strategy would be performed centrifugation technique with Plasma volume varying from 1.5 - 2.5 times the plasma - volume along with Standard Medical Treatment.
  Arms: Standard volume Therapeutic Plasma Exchange

SUMMARY:
In this prospective randomized controlled trial Investigator aim to evaluate the impact of high versus standard volume plasma-exchange in patients with acute liver failure with cerebral edema and clinical outcomes. ALF who meet the inclusion and exclusion criteria within the first 12 hours will be randomized into two groups

Interventional - High-volume plasma exchange Active Comparator - Standard volume plasma exchange

Expected outcome of the project-.

1. Primary end points: Time to improvement in cerebral edema
2. Secondary end points:

To study the adverse events of therapy (volume overload, pulmonary complications, allergic reactions) etc.

Transplant-free survival at day 21

DETAILED DESCRIPTION:
All patients will undergo plain CT-scan of the brain to screen for the presence and severity of cerebral edema in the emergency before being shifted to the L-ICU. In the L- ICU, patients will be managed by a multidisciplinary team. Intubation and ventilation will be undertaken for standard indications in addition to the development of grade 3 encephalopathy or evidence of cerebral edema on CT-scan. Ventilation will be managed by fentanyl and propofol along with the use of atracurium for paralysis wherever required. All patients will be monitored constantly for macro-hemodynamics, global tissue perfusion, and microcirculation. The macro-hemodynamic parameters included continuous monitoring of mean arterial pressure (MAP), heart rate and urine output per hour. The real-time monitoring of systemic vascular resistance (SVR), stroke volume variation (SVV), cardiac index (CI) and cardiac output (CO) will be done by a hemodynamic monitor (FloTrac™ system 4.0, Edwards Lifesciences, California, US) wherever feasible. Global tissue perfusion adequacy and indirect assessment of microcirculation will be done by measurement of arterial lactate. Fluid management will be done with crystalloids, with the use of colloids (5% albumin) in patients with severe hypoalbuminemia (serum albumin less than 2.5gm/dl). Norepinephrine will be the primary vasopressor used to target a mean arterial pressure of 65-70 mm of Hg. with adjunctive use of intravenous low dose hydrocortisone and vasopressin in patients not responsive to initial therapy.

Cerebral edema: The monitoring of cerebral edema will be performed measuring the optic nerve sheath diameter (ONSD) in both the eyes using a 7.5 MHz probe every 6-8 hours. Apart from this, routine monitoring of pupillary size and reactions, extensor posturing and plantar reflexes will be performed every 6-8 hrs. Transcranial doppler would be done every 6-8 hours. Patients will receive 3% hypertonic saline as a continuous infusion, initially started at 25ml /hr and titrated 6 hourly to between 5 and 20 mL per hour (maximum 100 ml/hour) to achieve serum sodium levels between 145-150 mmol/L. Intravenous 20% mannitol (1 g/kg IV bolus) over 20 to 30 minutes will be administered to those without renal failure. All patients will in addition receive intravenous N-acetylcysteine for 5 day.Routine electroencephalogram (EEG) will be done for all patients daily to screen for non-convulsive seizures which will be managed by intravenous levetiracetam. Assessment of coagulation will be performed by ROTEM at baseline and subsequently as required.

Protocol for therapeutic plasma-exchange TPE procedures will be performed using either Spectra Optia (SPO, Terumo BCT, Lakewood, CO, USA) continuous-flow centrifugal apheresis system or Haemonetics MCS+ (Braintree, MA, USA) intermittent flow centrifugal apheresis system via a double-lumen central venous dialysis catheter. All patients will receive plasma-exchange within first 12 hours of admission to the L-ICU along with a target volume of based on the randomization group per session. The replacement fluid used will be 90% FFP and 10% normal saline. TPE will be performed on consecutive days until the desired response is achieved. [using our previously published protocol].

The number of sessions of TPE in each patient will be decided based on the clinical response to SVPE. Dynamic assessment of the clinical parameters (signs of CE as assessed by pupillary size, reaction, and optic nerve-sheath diameter), INR, lactate and arterial ammonia will be performed at after each TPE. In patients with an improvement in INR, and signs of CE along with a reduction in ammonia at 6 hours which was sustained at 12 and 24 hours post-TPE, subsequent sessions will be discontinued. TPE will also be discontinued in patients who would show worsening in either clinical and/ or biochemical parameters. In patients who will develop adverse events, the TPE procedure will be resumed or discontinued depending on the severity of adverse event and its resolution. CRRT would be initiated in patients who develop worsening or ammonia or cerebral edema or metabolic complications and time to initiation of CRRT would be recorded in both groups. The time to initiation of CRRT would be recorded in both groups after randomization.

Continuous renal replacement therapy will be administered as continuous venovenous hemodiafiltration (CVVHDF) using Prisma and Prismaflex (Gambro) devices, with blood flows ranging from 150-180 mL/hr and target effluent rates of 20 - 25 mL/kg/hr. Anticoagulation was not used during dialysis. CRRT would be continued until resolution of cerebral edema and in decrease in ammonia levels below 150 ug/dl or in those who develop adverse effects of therapy.

Randomization will be done by taking 1:1 ratio by computer-generated sealed envelopes by the clinical trial co-ordinator.

Intervention group : High Volume PLsma Exchange (HVPE)+ Standard Medical Treatment (SMT) The high-volume strategy would be performed by centrifugation technique ~ 8-9 litres of plasma would be exchanged in each patient over 6-8 hours.

Active Comparator - The Standard volume Plasma Exchange + Standard medical Treatment The Standard volume strategy group Therapeutic Plasma Exchange would be performed varying from 1.5- 2.5 times the plasma - volume.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute liver failure defined as patients with jaundice which is complicated by encephalopathy and coagulopathy within 4 weeks of the onset of jaundice and without underlying chronic liver disease.

Cerebral edema documented on CT-scan and arterial ammonia >150 ug/dL

Exclusion Criteria:

1. Age <18 or > 70 years
2. HCC
3. Active untreated Sepsis/DIC
4. Hemodynamic instability non-responsive to initial fluid resuscitation with norepinephrine >0.1 ug/kg/min
5. Post-resection and malignancy related liver failure
6. Coma of non-hepatic origin
7. Patients with uncontrolled infection
8. Patients with pulmonary involvement with Pa02/Fio2 ratio below 200.
9. Patients with post renal obstructive AKI, AKI suspected due to glomerulonephritis, interstitial nephritis or vasculitis based on clinical history and urine analysis
10. Extremely moribund patients with an expected life expectancy of less than 24 hours
11. Pregnancy related liver failure
12. Comorbidities associated with poor outcome (Extrahepatic neoplasia, severe cardiopulmonary disease defined by a New York Heart Association score >3, or oxygen/steroid-dependent chronic obstructive pulmonary disease)
13. Refusal to participate in the study
14. Drug-induced ALF

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to improvement in cerebral edema | 7 Days
  Time to improvement in Cerebral Edema defined as sustained reduction in ammonia with resolution of Hepatic encephalopathy.

SECONDARY OUTCOMES:
To study the adverse events of therapy | 21 Days
  Adverse Events- Pulmonary complications, allergic reactions, hypotension, etc
Transplant-free survival at day 21 | 21st day
  Time to death and liver transplant will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 Month